CLINICAL TRIAL: NCT07252817
Title: Seguimiento Intensivo Del Dolor Postoperatorio en cirugía Mayor Ambulatoria: Estudio de Viabilidad y Resultados
Brief Title: Intensive Monitoring of Post-surgery Pain in Major Ambulatory Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari del Maresme (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIm04/25
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Hernioplasty; Cholecystectomy, Laparoscopic; Haemorrhoidal Surgery; Knee Arthroscopy; Shoulder Arthroscopy
Keywords: Pain; Post-surgery pain; pain control
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard monitoring group (Active Comparator): Routine follow-up (telephone call on the morning after surgery)
  Interventions: Other: Standard monitoring group
- Intensive monitoring group (Experimental): Routine follow-up (telephone call on the morning after surgery) and Intensive follow-up of acute post-surgery pain.
  Interventions: Other: Intensive monioring group

INTERVENTIONS:
Other: Intensive monioring group — Routine follow-up (telephone call on the morning after surgery) and Intensive follow-up of acute post-surgery pain (telephone call every day since pain resolution).
  Arms: Intensive monitoring group
Other: Standard monitoring group — Routine follow-up (telephone call on the morning after surgery).
  Arms: Standard monitoring group

SUMMARY:
Moderate to severe acute postoperative pain (APP) during part of the postoperative period is a barrier that hinders the central objective of perioperative medicine, which is to achieve an optimal postoperative recovery process. Despite advances in perioperative medicine, a large proportion of post-operative patients continue to suffer from moderate to severe APS during many of the days of their convalescence. This poor control of APS, in addition to causing suffering and exposing the patient to an increased risk of complications, could impair the quality of post-surgical recovery , according to some authors. We therefore consider it to be of utmost interest in our field to corroborate whether the implementation of measures to better control DAP is related to a better quality of post-surgical recovery.

Currently, the growing trend to take into account the perspective of patients in their care has prompted the development of various patient-centred measurement tools that, among other aspects, assess the quality of post-surgical recovery. Several scales have been designed. The most widely used are the QoR-40, QoR-9 and QoR-15 scales. The latter, with a range of 0 to 150, was developed to simplify assessment, especially in telephone follow-ups, and has a reliability similar to its predecessor, the QoR-40.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old.
* ASA I - III.
* Scheduled for the surgeries: Laparoscopic or open inguinal hernia repairs, Laparoscopic cholecystectomies, Haemorrhoid surgeries, Knee arthroscopies, Shoulder arthroscopies.
* Willingness to be contacted by telephone during the duration of the study.
* Informed written consent to participate in this study.

Exclusion Criteria:

* Lack of proficiency in Spanish.
* Undergoing study or follow-up for moderate to severe cognitive impairment.
* Pregnant or breastfeeding patients.
* Patients on major opioid medication.
* Patients with a history of dependence/abuse of alcohol or illicit drugs at present.
* Patients under active follow-up by the chronic pain unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery | Baseline (pre-surgery) and 48 hours, 7 days and 14 days post-surgery
  Quality of Recovery (QoR15 test)

SECONDARY OUTCOMES:
Pain Control by Visual Analogic Scale | Baseline (pre-surgery) and 48 hours, 7 days and 14 days post-surgery
  Visual Analogic Scale of pain. Range values: 0 (minium pain) thru 10 (maximum pain)
Satisfaction of pain control | Baseline (pre-surgery) and 48 hours, 7 days and 14 days post-surgery
  A 4-level Likert scale will be used according to the patient's criteria: dissatisfied, slightly dissatisfied, fairly satisfied, completely satisfied.
Adherence to prescribed analgesic treatment | Baseline (pre-surgery) and 48 hours, 7 days and 14 days post-surgery
  4-level Likert scale according to the patient's criteria: no adherence, low adherence, moderate adherence, and total adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Sanitari del Maresme, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No